CLINICAL TRIAL: NCT01431235
Title: Investigating the Efficacy of Cognitive Behavioral Therapy in Patients With Substance Use Disorder and Comorbid ADHD. A Randomized Controlled Trial With Cognitive Behavioral Therapy
Brief Title: CBT for Patients With Attention Deficit Hyperactivity Disorder (ADHD) and Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkin (Industry)
Collaborators: Fonds NutsOhra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-130
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Attention Deficit Hyperactivity Disorder; Substance Use Disorders
Keywords: ADHD; SUD; cognitive behavioral therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard addiction treatment (No Intervention): 10 sessions of standard addiction treatment. No ADHD treatment.
- addiction treatment and ADHD treatment (Experimental): 10 sessions cognitive behavioral therapy on addiction treatment combined with 5 sessions on ADHD treatment.
  Interventions: Behavioral: cognitive behavioral therapy for treating ADHD symptoms

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for treating ADHD symptoms — 5 sessions of one hour CBT for treating ADHD symptoms by a trained health care worker
  Arms: addiction treatment and ADHD treatment

SUMMARY:
The purpose of this study is to determine if cognitive behavioral therapy is effective in treating ADHD symptoms in patients with substance use disorders and comorbid ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder(ADHD) is an important comorbid condition in patients with substance use disorders (SUD). The prevalence of ADHD in patients with SUD is estimated 23%, and ADHD is associated with an untoward prognosis of SUD. However, adequate treatment programs for patients with ADHD and SUD are not available. Results of medication trials for patients with ADHD and SUD are disappointing, and cognitive behavioral therapy (CBT) has not yet been investigated in this population. In patients with ADHD without comorbid SUD, the results of CBT in randomized trials are positive. The purpose of this study is to investigate if CBT is effective in treating ADHD symptoms in patients with ADHD and SUD.

ELIGIBILITY:
Inclusion Criteria:

* substance use disorder
* ADHD
* able to comply with study activities

Exclusion Criteria:

* severe neurological or psychiatric diseases (for example Parkinson, dementia, psychosis, bipolar depression) which require medication
* unable to read or write Dutch language

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
self reported ADHD symptoms | 6 months
  Dutch self report list of ADHD symptoms by Kooij and Buitelaar

SECONDARY OUTCOMES:
Time Line Follow Back method | 6 months
  self-reported alcohol and drug use
Beck depression inventory | 6 months
  self reported depression symptoms
Beck Anxiety Inventory | 6 months
  Self reported anxiety symptoms
EQ-5 | 6 months
  Self reported quality of living
TIC-P | 6 months
  health care consumption and production loss in relation to mental health problems
Stroop task | 6 months
  neuropsychological measure
Tower of London task | 6 months
  neuropsychological task
BART task | 6 months
  neuropsychological task on risk taking behavior
urine checks | 6 months
  urine checks on drug use

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schoevers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Arkin, Amsterdam, Netherlands

REFERENCES:
- [Background] Arias AJ, Gelernter J, Chan G, Weiss RD, Brady KT, Farrer L, Kranzler HR. Correlates of co-occurring ADHD in drug-dependent subjects: prevalence and features of substance dependence and psychiatric disorders. Addict Behav. 2008 Sep;33(9):1199-207. doi: 10.1016/j.addbeh.2008.05.003. Epub 2008 May 13. PMID 18558465
- [Background] Castells X, Ramos-Quiroga JA, Rigau D, Bosch R, Nogueira M, Vidal X, Casas M. Efficacy of methylphenidate for adults with attention-deficit hyperactivity disorder: a meta-regression analysis. CNS Drugs. 2011 Feb;25(2):157-69. doi: 10.2165/11539440-000000000-00000. PMID 21254791
- [Background] Safren SA, Sprich S, Mimiaga MJ, Surman C, Knouse L, Groves M, Otto MW. Cognitive behavioral therapy vs relaxation with educational support for medication-treated adults with ADHD and persistent symptoms: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):875-80. doi: 10.1001/jama.2010.1192. PMID 20736471
- [Background] Solanto MV, Marks DJ, Wasserstein J, Mitchell K, Abikoff H, Alvir JM, Kofman MD. Efficacy of meta-cognitive therapy for adult ADHD. Am J Psychiatry. 2010 Aug;167(8):958-68. doi: 10.1176/appi.ajp.2009.09081123. Epub 2010 Mar 15. PMID 20231319
- [Derived] van Emmerik-van Oortmerssen K, Vedel E, Koeter MW, de Bruijn K, Dekker JJ, van den Brink W, Schoevers RA. Investigating the efficacy of integrated cognitive behavioral therapy for adult treatment seeking substance use disorder patients with comorbid ADHD: study protocol of a randomized controlled trial. BMC Psychiatry. 2013 May 10;13:132. doi: 10.1186/1471-244X-13-132. PMID 23663651